CLINICAL TRIAL: NCT06152393
Title: Retro-prospective Multicentric Study Aiming to Evaluate the Benefit of Measuring an Intrathecal Synthesis Index of Specific Antitreponema IgG for Patients Suspected of Neurosyphilis
Brief Title: Value of an Intrathecal Synthesis Index of Specific Antitreponema IgG for Neurosyphilis Diagnosis
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: Swiss HIV Cohort Study (Network); Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Laurence Toutous Trellu, Principal Investigator, University Hospital, Geneva
Other Study IDs: Study 2019-00232
Record Dates: First submitted 2023-10-12; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Neurosyphilis
Keywords: Neurosyphilis; Treponema pallidum; Intrathecal synthesis; Specific anti-Treponema IgG; Otosyphilis; Ocular syphilis
MeSH Terms: conditions — Neurosyphilis; Treponemal Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control patients: Controls were patients diagnosed with TPHA/TPPA serology ≥80 and neurological symptoms requiring a lumbar puncture.
  Interventions: Diagnostic Test: Measure of an antibody index for intrathecal synthesis of specific anti-Treponema pallidum IgG by ELISA.
- NS1 patients: NS1 includes: 1) neurological symptoms suggestive of central nervous system (CNS) involvement or acute ophthalmological or acute auditory signs consistent with neurosyhilis (NS), or syphilis with treatment serological failure (< fourfold decrease in the antibody titer of RPR/VDRL 12 months after treatment), and 2) a TPHA/TPPA serology ≥ 80 and a CSF-TPHA/TPPA test ≥ 320, and 3) either CSF-WBC > 5 cells/mm3, and/or CSF-protein > 0,45g/l in the absence of other known causes of these abnormalities, and/or a reactive CSF-VDRL/RPR test, and 4) no differential diagnosis.
  Interventions: Diagnostic Test: Measure of an antibody index for intrathecal synthesis of specific anti-Treponema pallidum IgG by ELISA.
- NS2 patients: NS2 includes:1) acute ocular symptoms (recent and sudden decrease in visual acuity) and/or acute otologic dysfunctions (sudden hearing loss, acute tinnitus or vertigo) without other known diagnosis for these clinical abnormalities, 2) and a TPHA/TPPA serology ≥ 80, 3) and a response to NS treatment assessed by ophthalmologic or hearing tests and at least a fourfold reduction of RPR/VDRL titer in blood after 12 months following treatment.
  Interventions: Diagnostic Test: Measure of an antibody index for intrathecal synthesis of specific anti-Treponema pallidum IgG by ELISA.

INTERVENTIONS:
Diagnostic Test: Measure of an antibody index for intrathecal synthesis of specific anti-Treponema pallidum IgG by ELISA. — Paired CSF/serum samples from all patients were blind tested for anti-T. pallidum IgG with an ELISA containing recombinant T. pallidum proteins (Euroimmun).
  The AI was calculated conforming to Reiber's method (PMID 11239944) and as previously described in Alberto et al. (PMID 35138118).

SUMMARY:
A retro-prospective case-control Swiss study was conducted to evaluate the diagnostic performance of measuring an antibody index (AI) for intrathecal synthesis of specific anti-Treponema pallidum (T. pallidum) IgG for the diagnosis of neurosyphilis.

DETAILED DESCRIPTION:
The diagnosis of neurosyphilis (NS) lacks a true "gold standard" which makes the diagnosis challenging while consequences of a misdiagnosis are potentially severe. The aim of this study was to evaluate the diagnostic performance of measuring an antibody index (AI) for intrathecal synthesis of specific anti-Treponema pallidum (T. pallidum) IgG for the diagnosis of NS.

CSF parameters were analysed and specific anti-T. pallidum IgG were measured simultaneously on paired cerebrospinal fluid (CSF)-serum samples collected between 2007 and 2022 from patients suspected of NS, in Switzerland. An AI was calculated to consider blood-brain barrier integrity. Two NS definitions were used: NS1 included patients with suspicion of NS presenting neurological symptoms and/or acute neuro-sensory signs and positive TPHA/TPPA serology and CSF-TPHA/TPPA≥320, and either CSF-leucocytes >5cells/mm3 and/or CSF-protein >0,45g/l and/or a reactive CSF-VDRL/RPR test. NS2 included patients with NS suspicion presenting acute ocular and/or otologic symptoms, and positive TPHA/TPPA serology, and a favourable response to NS treatment. Controls were patients diagnosed with any other CNS pathologies and with positive TPHA/TPPA serology.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have serum / CSF sample pairs collected concomitantly (3 days maximum interval between blood test and lumbar puncture).
* Age > or = 18 years old.

Exclusion Criteria:

* All patients for whom the stored samples do not meet the needs of the diagnostic study, or whose serum and CSF collection date is more than 3 consecutive days.
* Age < 18 years old.
* No written consent form for the prospective part.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a bidirectional retrospective and prospective multicenter study, including all the patients presenting neurological and neuro-sensory signs (ophthalmic and auditory), for whom we have serum and cerebrospinal fluid samples, from the University Hospitals of Geneva, Zurich and Lausanne, at the ADMED Microbiology Laboratory of La Chaux-de-Fonds and in SHCS centers.
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of the diagnostic performance of measuring an antibody index (AI) for intrathecal synthesis of specific anti-Treponema pallidum IgG for the diagnosis of neurosyphilis. | 2020-2022 with retrospective samples from 2007 to 2019 and prospective samples from 2019 to 2022.
  AI testing measured with an Elisa specific for anti-Treponema pallidum IgG for all patients : number of patients with positive AI, sensitivity/specificity of the test, and positive/negative predictive values of AI test were estimated.

SECONDARY OUTCOMES:
Intrathecal oligoclonal IgG production analysis | 2020-2022 with retrospective samples from 2007 to 2019 and prospective samples from 2019 to 2022.
  IgG oligoclonal bands were analysed in CSF and serum of NS and control patients by the gold standard isoelectric focusing method

CONTACTS AND LOCATIONS:
Locations (1):
- Laurence Toutous Trellu, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reiber H, Peter JB. Cerebrospinal fluid analysis: disease-related data patterns and evaluation programs. J Neurol Sci. 2001 Mar 1;184(2):101-22. doi: 10.1016/s0022-510x(00)00501-3. PMID 11239944
- [Background] Alberto C, Deffert C, Lambeng N, Breville G, Gayet-Ageron A, Lalive P, Toutous Trellu L, Fontao L. Intrathecal Synthesis Index of Specific Anti-Treponema IgG: a New Tool for the Diagnosis of Neurosyphilis. Microbiol Spectr. 2022 Feb 23;10(1):e0147721. doi: 10.1128/spectrum.01477-21. Epub 2022 Feb 9. PMID 35138118